CLINICAL TRIAL: NCT04991766
Title: An Open-label, Two-part Study of the Disposition and Absolute Bioavailability of [¹⁴C]-LY3484356 in Healthy Females of Non-Childbearing Potential
Brief Title: A Study of [¹⁴C]-LY3484356 in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18205; J2J-MC-JZLE (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-08-02; First posted 2021-08-05 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11-15

CONDITIONS: Healthy
Keywords: Metabolism; Absolute Bioavailability; Disposition
MeSH Terms: interventions — Imlunestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [¹⁴C]-LY3484356 (Part 1) (Experimental): Participants received a single oral dose of 400 mg Carbon 14 labelled [¹⁴C]-LY3484356 following an overnight fast of at least 10 hours on Day 1.
  Interventions: Drug: [¹⁴C]-LY3484356
- LY3484356 + [¹⁴C]-LY3484356 (Part 2) (Experimental): Participants received a single oral dose of 400 mg LY3484356 following an overnight fast of at least 10 hours on Day 1, followed 4 hours later by a single dose of less than 100 microgram (μg) [¹⁴C]-LY3484356 (actual ranged from 44.55 to 45.95 μg), as an intravenous (IV) infusion on day 1.
  Interventions: Drug: LY3484356; Drug: [¹⁴C]-LY3484356 (IV)

INTERVENTIONS:
Drug: [¹⁴C]-LY3484356 — Administered orally.
  Arms: [¹⁴C]-LY3484356 (Part 1)
Drug: LY3484356 — Administered orally.
  Arms: LY3484356 + [¹⁴C]-LY3484356 (Part 2)
Drug: [¹⁴C]-LY3484356 (IV) — Administered IV.
  Arms: LY3484356 + [¹⁴C]-LY3484356 (Part 2)

SUMMARY:
The main purpose of this study is to measure how much of the study drug gets into the bloodstream and how long it takes the body to get rid of it. This study has two parts. It will involve a single dose of 14C radiolabeled LY3484356. This means that a radioactive substance C14 will be incorporated into the study drug, to investigate the study drug and its breakdown products, to find out how much of these pass from blood into urine, feces and expired air. The study will last about 4 weeks. Screening is required within 28 days prior to the start of the study and follow up is required approximately 7 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of nonchildbearing potential. This includes females who are not pregnant, non-lactating and either: Infertile due to surgical sterilization or alternate medical cause/congenital or postmenopausal.
* Body mass index (BMI) within the range of 18.0 to 35.0 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorders
* Have evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Have known allergies to LY3484356, related compounds or any components of the formulation as appropriate, or history of significant atopy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LabCorp CRU, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a two-part study. Participants in Part 1 did not participate in Part 2.
Groups:
- Part 1: [¹⁴C]-LY3484356: Participants received a single oral dose of 400 milligram (mg) Carbon 14 labelled [¹⁴C]-LY3484356 following an overnight fast of at least 10 hours on Day 1.
- Part 2: LY3484356 + [¹⁴C] LY3484356: Participants received a single oral dose of 400 mg LY3484356 following an overnight fast of at least 10 hours on Day 1, followed 4 hours later by a single dose of less than 100 microgram (μg) [¹⁴C]-LY3484356 (actual ranged from 44.55 to 45.95 μg), as an intravenous (IV) infusion on day 1.
Period: Overall Study
Arm/Group | Part 1: [¹⁴C]-LY3484356 | Part 2: LY3484356 + [¹⁴C] LY3484356
Started | 8 | 8
Received at Least 1 Dose of Study Drug | 8 | 8
Completed | 6 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug (LY3484356 or [¹⁴C]-LY3484356).
Groups:
- Part 1: [¹⁴C]-LY3484356: Participants received a single oral dose of 400 mg Carbon 14 labelled [¹⁴C]-LY3484356 following an overnight fast of at least 10 hours on Day 1.
- Part 2: LY3484356 + [¹⁴C] LY3484356: Participants received a single oral dose of 400 mg LY3484356 following an overnight fast of at least 10 hours on Day 1, followed 4 hours later by a single dose of less than 100 μg [¹⁴C]-LY3484356 (actual ranged from 44.55 to 45.95 μg), as an IV infusion on day 1.
- Total: Total of all reporting groups
Arm/Group | Part 1: [¹⁴C]-LY3484356 | Part 2: LY3484356 + [¹⁴C] LY3484356 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (7.1) | 53.3 (9.4) | 53.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 3 | 5 | 8
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Pharmacokinetics (PK): Fecal Excretion of LY3484356 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: The percentage of the total radioactive dose administered that was excreted in feces = (amount of radioactive dose recovered in feces / total radioactive dose administered) * 100.
Time Frame: Predose, 24, 48, 72, 96, 120, 144, 168,192, 216, 240, 264, 288 and 312 hours post dose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Mean (Full Range); unit: percentage of the total radioactive dose
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 5
percentage of the total radioactive dose | 97.3 [90.0 to 101.0]

2. Primary Outcome: Part 1: PK: Urinary Excretion of LY3484356 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: The percentage of the total radioactive dose administered that was excreted in urine = (amount of radioactive dose recovered in urine / total radioactive dose administered) * 100.
Time Frame: Predose, 24, 48 ,72, 96, 120, 144, 168, 192, 216, 240, 264, 288 and 312 hours post dose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Mean (Full Range); unit: percentage of the total radioactive dose
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 5
percentage of the total radioactive dose | 0.278 [0.109 to 0.497]

3. Primary Outcome: Part 2: Pharmacokinetics (PK): Percent Absolute Bioavailability (F%) of LY3484356
Description: PK: Bioavailability is defined as the percentage of a drug which enters the circulation when introduced into the body and so is able to have an active effect. Percent absolute bioavailability, calculated for plasma LY3484356 as "F %= [AUC (0-∞), LY3484356] × [Dose, [14C]-LY3484356] / [AUC (0-∞), [14C]-LY3484356] × [Dose, LY3484356] ×100%'' Higher percent indicates better absorption of drug into the body.
Time Frame: Predose, 5 minutes(min), 15 min, 20 min, 30 min, 45 min, and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours postdose
Population: All enrolled participants who received at least 1 dose of LY3484356 + [¹⁴C]-LY3484356 and have evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent absolute bioavailability
Groups:
- Part 2: LY3484356 + [¹⁴C]-LY3484356: Participants received a single oral dose of 400 mg LY3484356 following an overnight fast of at least 10 hours on Day 1, followed 4 hours later by a single dose of less than 100 μg [¹⁴C]-LY3484356 (actual ranged from 44.55 to 45.95 μg) as an IV infusion on day 1.
Arm/Group | Part 2: LY3484356 + [¹⁴C]-LY3484356
Number analyzed (Participants) | 8
percent absolute bioavailability | 10.5 (32)

4. Secondary Outcome: Part 1: PK: Total Radioactivity Recovered in Urine, Feces
Description: Relative abundance was expressed and calculated as the percentage of administered dose excreted in urine/Feces=[(percentage of radioactivity in peak)/100]*(percentage of dose in sample).
Time Frame: Predose, 24, 48, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456 and 480 hours post dose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Mean (Full Range); unit: percentage of recovered radioactivity
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 5
percentage of recovered radioactivity
  Urine Radioactivity | 0.278 [0.109 to 0.497]
  Fecal Radioactivity | 97.3 [90.0 to 101.0]

5. Secondary Outcome: Part 1: Total Radioactivity Recovered in Expired Air
Description: Radioactivity is expressed in becquerels (Bq), the International System of Unit (SI) representing one nuclear disintegration per second. For practical measurement, total radioactivity recovered in expired air is reported in disintegrations per minute (dpm). The conversion factor is: 1 Bq = 60 dpm.
Time Frame: predose, 8, and 24 hours postdose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Number; unit: disintegrations per minute
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 1
disintegrations per minute
  8 hours postdose | 53
  24 hours postdose | 62

6. Secondary Outcome: Part 1: PK: Total Number of Metabolites of LY3484356 in Plasma, Urine and Feces
Description: Total number of metabolites of LY3484356 is reported. The value is an absolute number without any measure of central tendency.
Time Frame: Plasma:Predose,24,48,72,96,120,144,168,192,216,240,264 and 288 hours(h) post dose;Urine:-12 to 0h Predose,0 to 6,6-12,and 12-24,48,72,96,120,144,168,192,216,240 and 264 hours post dose;Feces:Predose,24,48,72,96,120,144, 168,192,216,240 and 264 h post dose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Number; unit: number of metabolites
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 5
number of metabolites
  Plasma | 3
  Urine | 0
  Feces | 7

7. Secondary Outcome: Part 1: PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC [0-∞]) for LY3484356 in Plasma
Description: PK: AUC [0-∞] of LY3484356 in Plasma.
Time Frame: Part 1: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8,10, 12, 24, 48, 72, 96,120, 144, 168, 192, 216, 240, and 264 hours post-dose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 6
nanogram*hour per milliliter (ng*hr/mL) | 3130 (38)

8. Secondary Outcome: Part 1: PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC [0-∞]) for Total Radioactivity in Plasma
Description: PK: AUC [0-∞] of Plasma Total Radioactivity.
  Total radioactivity is reported as nanogram* hours equivalents per milliliter (ng*h Eq/mL).
Time Frame: as for outcome 7
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h Eq/mL
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 6
ng*h Eq/mL | 17900 (39)

9. Secondary Outcome: Part 1: PK: Maximum Concentration (Cmax) for LY3484356 in Plasma
Description: PK: Cmax for LY3484356 in plasma.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8,10, 12, 24, 48, 72, 96,120, 144, 168, 192, 216, 240, and 264 hours post-dose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL) | 108 (48)

10. Secondary Outcome: Part 1: PK: Maximum Concentration (Cmax) for Total Radioactivity in Plasma
Description: PK: Cmax for total radioactivity in plasma. The Cmax of total radioactivity are reported as nanogram equivalents per milliliter (ng Eq/mL).
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8,10, 12, 24, 48, 72, 96,120, 144, 168, 192, 216, 240, and 264 hours post-dose
Population: All enrolled participants who received at least 1 dose of [¹⁴C]-LY3484356 and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq/mL
Arm/Group | Part 1: [¹⁴C]-LY3484356
Number analyzed (Participants) | 6
ng Eq/mL | 537 (18)

11. Secondary Outcome: Part 2: PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC [0-∞]) for [¹⁴C]-LY3484356 and LY3484356 in Plasma
Description: PK: AUC [0-∞] of Total Radioactivity.
  Total radioactivity is reported as hours*nanogram equivalents per milliliter (h*ng Eq/mL).
Time Frame: as for outcome 3
Population: All enrolled participants who received at least 1 dose of LY3484356 or [¹⁴C]-LY3484356 and have evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: LY3484356 + [¹⁴C]-LY3484356
Number analyzed (Participants) | 8
ng*hr/mL
  Plasma [14C]-LY3484356 | 1.95 (26)
  Plasma LY3484356 | 1810 (45)

12. Secondary Outcome: Part 2: PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC [0-∞]) for Total Radioactivity in Plasma
Description: PK: AUC [0-∞] of Total Radioactivity in Plasma.
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h Eq/mL
Arm/Group | Part 2: LY3484356 + [¹⁴C]-LY3484356
Number analyzed (Participants) | 8
ng*h Eq/mL | 7.44 (18)

13. Secondary Outcome: Part 2: PK: Maximum Concentration (Cmax) for [¹⁴C]-LY3484356 and LY3484356 in Plasma
Description: PK: Cmax of LY3484356 and [¹⁴C]-LY3484356 in plasma.
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: LY3484356 + [¹⁴C]-LY3484356
Number analyzed (Participants) | 8
ng/mL
  Plasma [14C]-LY3484356 | 0.575 (21)
  Plasma LY3484356 | 33.1 (59)

14. Secondary Outcome: Part 2: PK: Maximum Concentration (Cmax) for Total Radioactivity in Plasma
Description: PK: Cmax of total radioactivity in plasma.
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq/mL
Arm/Group | Part 2: LY3484356 + [¹⁴C]-LY3484356
Number analyzed (Participants) | 8
ng Eq/mL | 0.857 (18)

ADVERSE EVENTS:
Time Frame: Part 1: Baseline Up to Day 29, Part 2: Baseline Up to Day 16
Description: All enrolled participants who received at least 1 dose of LY3484356 or [14C]-LY3484356, whether or not they completed all protocol requirements.
Groups:
- Part 2: LY3484356 + [¹⁴C]-LY3484356: Participants received a single oral dose of 400 mg LY3484356 following an overnight fast of at least 10 hours on Day 1, followed 4 hours later by a single dose of less than 100 μg [¹⁴C]-LY3484356 (actual ranged from 44.55 to 45.95 μg), as an IV infusion on day 1.
Arm/Group | Part 1: [¹⁴C]-LY3484356 | Part 2: LY3484356 + [¹⁴C]-LY3484356
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: [¹⁴C]-LY3484356 (N=8) | Part 2: LY3484356 + [¹⁴C]-LY3484356 (N=8)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04991766/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT04991766/SAP_001.pdf